CLINICAL TRIAL: NCT04586842
Title: Study Protocol For A Non-Randomised Controlled Trial: A Community-Based Occupational Therapy Intervention On Mental Health For People With Acquired Brain Injury (COT-MHABI)
Brief Title: Community-based Occupational Therapy Intervention on Mental Health for People With Acquired Brain Injury
Acronym: COT-MHABI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Guttmann (Other)
Collaborators: University of Vic - Central University of Catalonia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 252136
Record Dates: First submitted 2020-07-21; First posted 2020-10-14 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Acquired Brain Injury; Mental Health Issue
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community-based Occupational Therapy (Experimental): Experimental study group that will receive a domiciliary and community-based occupational therapy on mental health, developed on the basis of the Model Of Human Occupation.
  Interventions: Behavioral: Community-based Occupational Therapy
- Standard community-based intervention (Active Comparator): Control group of the study that will receive community-based interventions, public or private level (e.g. community nursing, social education and/or psychology).
  Interventions: Behavioral: Standard community-based intervention

INTERVENTIONS:
Behavioral: Community-based Occupational Therapy — Domiciliary and Community-based Occupational Therapy on mental health and ABI intervention, developed on the basis of the Model Of Human Occupation.
  Arms: Community-based Occupational Therapy
Behavioral: Standard community-based intervention — Interventions received at the community, public or private level (e.g. community nursing, social education and/or psychology).
  Arms: Standard community-based intervention

SUMMARY:
The main purpose of this research project is to analyze the effectiveness of a Community-based Occupational Therapy Intervention on mental health for people with acquired brain injury. To this end, variables such as quality of life, occupational performance and balance, participation in significant roles and community integration will be measured.

The research will be carried out as a non-randomized controlled trial study in which the participants in the experimental arm will receive a community-based occupational therapy intervention (domiciliary and telehealth intervention sessions) based on the stages of the Human Occupation Model's Remotivation Process. The participants at the control arm will receive the regular (public or private) services provision for this population profile.

It is expected to be able to demonstrate the effectiveness of the intervention based on a positive result in the change in the variables, so as to increase the chance and performance of occupational participation after the acquired brain injury. Also, it is intended that families and the community are key elements of agency and support in occupational participation.

ELIGIBILITY:
Inclusion criteria:

Adults with a diagnosis of medium or severe ABI and a diagnosis of neurocognitive disorder following ABI (as recognised in the 5th edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5); by definition: evidence of significant cognitive decline from pre-ABI level in one or more cognitive domains (attention, executive function, learning and memory, perceptual-motor ability or social cognition).

It may occur with or without behavioural impairment (apathy, mood disturbance, irritability, disinhibition, psychotic symptoms, etc.)).

This population (A) show difficulties in occupational participation with respect to the pre-ABI situation and present needs for support, counselling and/or specific therapeutic intervention; (B) are in a situation of hospital discharge from ABI specialisation units; (C) are domiciled in the same province to which the providing hospital belongs. In addition, they may or may not have been diagnosed with a mental health disorder other than neurocognitive disorder, either prior or subsequent to the ABI.

Exclusion criteria:

Persons will be excluded if (A) they are in a situation of symptomatological destabilisation of severe functional impairment that, as a priority, requires continued support from specialised mental health units, psychiatric or social-health care admission; and/or (B) they are unable to determine for themselves (for cognitive reasons or by conscious choice) any problem in at least one occupational area.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
World Health Organization Quality of Life-BREF, spanish version (WHOQoL-BREF) | 1 year
  This scale provides a profile of quality of life perceived by the subject.
Canadian Occupational Performance Measure, spanish version (COPM) | 1 year
  This scale is an evidence-based outcome measure designed to capture a client's self-perception of performance in everyday living, over time.

SECONDARY OUTCOMES:
Community Integration Questionnaire, spanish version (CIQ) | 1 year
  Provides the measure of an individual's level of integration into the home and community following traumatic brain injury.
Activity Card Sort, spanish version (ACS) | 1 year
  An Occupational Therapy scale that measures the level of participation perceived by the person through the use of photographs that reflect everyday activities.
Satisfaction with Daily Occupations and Occupational Balance, spanish version (SOD-EO) | 1 year
  An occupational therapy measure that provides information about the activity level of the subject, occupational satisfaction with his/her performance and self-perception of occupational balance.
Role Checklist Version 3 (RCV3) | 1 year
  An occupational therapy measure that provides information about the participation and satisfaction with performance in desired and meaningful roles.
Functional Independence Measure (FIM) | 1 year
  The scale represents a uniform measurement system for functional independence based on the International Classification of Impairment, Disabilities and Handicaps. It assesses six functional areas (self-care, sphincter control, transfers, locomotion, communication and social cognition) within two domains (motor and cognitive). Each item is scored on a 7-point Likert-type scale. The items are performance-based rather than ability-based and are recorded in a hetero-administered manner.

CONTACTS AND LOCATIONS:
Overall Officials: José A Merchán-Baeza, Study Director — University of Vic-UCC
Locations (1):
- Institut Guttmann Neurorehabilitation Hospital, Badalona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Raya-Ruiz MA, Rodriguez-Bailon M, Castano-Monsalve B, Vidana-Moya L, Fernandez-Solano AJ, Merchan-Baeza JA. Study protocol for a non-randomised controlled trial: Community-based occupational therapy intervention on mental health for people with acquired brain injury (COT-MHABI). PLoS One. 2022 Oct 7;17(10):e0274193. doi: 10.1371/journal.pone.0274193. eCollection 2022. PMID 36206208